CLINICAL TRIAL: NCT05433935
Title: A Prospective, Open Large Cohort Study of Intraductal Papillary Mucinous Neoplasm (IPMN) of the Pancreas
Brief Title: Exploring Biomarkers of the Carcinogenesis of Intraductal Papillary Mucinous Neoplasm (IPMN) of the Pancreas
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang, Zhejiang University
Other Study IDs: PCIPMN
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Intraductal Papillary Mucinous Neoplasm
Keywords: intraductal papillary mucinous neoplasm; biomarkers; prospective cohort
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The fresh blood, urine, feces and saliva of each patient will be collected during the surveillance. The samples of each patient will be collected at the following time points: 1) at diagnosis time of IPMN; 2) every 6 months during surveillance until malignant transformation. If patients receive surgical resection for targeted lesions, surgical specimens will also be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective IPMN cohort: Multi-omics analysis of 5000 prospectively collected samples.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This is an observational study.

SUMMARY:
This is a prospective, open large cohort study to explore biomarkers for detecting early carcinogenesis of IPMN.

DETAILED DESCRIPTION:
This prospective study was designed to explore biomarkers for detecting early carcinogenesis of IPMN. This study intends to prospectively and continuously enroll IPMN patients, and regularly collect biological samples including blood, urine, feces and saliva. We aimed to detect biomarkers which can predict the carcinogenesis of IPMN by multi-omics. The primary endpoint is the predictive accuracy of biomarkers for IPMN malignant transformation. The probability of IPMN malignant transformation , rates of surgical resection and survival after surgery are secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as IPMN;
* without other malignant tumor;
* agree to sign informed consent.

Exclusion Criteria:

* with mental disorders which can affect cognition and cooperation;
* with serious blood diseases or taking drugs that can affect peripheral blood

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients ought to meet all inclusion and exclusion criteria. In addition, the patient of the prospective cohort should be thoroughly informed about the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent of the prospective cohort should be obtained from the patient prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of IPMN malignant transformation | Up to 10 years

SECONDARY OUTCOMES:
the probability of IPMN malignant transformation | Up to 10 years
rates of surgical resection | Up to 10 years
survival after surgery | Up to 10-15 years

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, PhD, Study Chair — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No